CLINICAL TRIAL: NCT04610359
Title: Safety of Human Embryonic Stem Cell (hESC)-Derived Mesenchymal Stem Cells in Interstitial Cystitis; Open-labelled, Single Center, Phase 1 Study
Brief Title: Safety of Human Embryonic Stem Cell (hESC)-Derived Mesenchymal Stem Cells in Interstitial Cystitis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: MIRAE CELL BIO (Unknown)
Responsible Party: Principal Investigator, Myung-Soo Choo, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1451
Record Dates: First submitted 2020-10-19; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Interstitial Cystitis; Stem Cell Transplant; Mesenchymal Stem Cell
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stem cell group (Experimental): Interstitial cystitis patients who receive submucosal injection of hESC-MSCs
  Interventions: Drug: MR-MC-01

INTERVENTIONS:
Drug: MR-MC-01 — Submucosal injection of 2.0 x 10,000,000/5ml (1mL * 5 sites)

SUMMARY:
This study primarily aimed to evaluate the safety of human embryonic stem cell (hESC)-derived mesenchyma stem cells in interstitial cystitis.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged >= 20 years
* Interstitial cystitis symptom duration more than 6 months
* Presence of Hunner lesions in outpatient cystoscopy (within one months of screening), with size < 2cm, number <= 2
* VAS (Visual pain analogue scale) >=4 in screening symptom questionnaire
* Those who are suitable for stem cell transplantation

  * normal laboratory findings (hematological, chemical)
  * no history of drug abuse
  * negative HIV, HBV, HCV serology tests
  * No history of malignancies
  * willing to contraception
  * no plan for blood, tissue donation
* Who can understand consent form and willing to participate in the study

Exclusion Criteria:

* recurrent urinary tract infection ( more than twice per past six months or more than three times per past one year) or active urinary tract infection
* any active or past history of tuberculosis or systemic infection
* Anatomical abnormality of lower urinary tract
* History of following procedures

  * stem cell transplantation In past 6 months,
  * transurethral resection/fulguration of Hunner lesion or hydrodistension of bladder
  * intravesical instillation of ialuril
  * hysterectomy, anti-incontinence surgery, transvaginal surgery, pelvic organ prolapse repair, vagina delivery or C/sec
  * any neurological conditions including cerebrovascular disease, multiple sclerosis, spinal cord injury, Parkinson disease
  * indwelling Foley catheter or intermittent catheterization
  * any plans for electrostimulation, neuromodulation, physiotherapy or operation for other organs
  * any history of malignancy
  * history of myocardiac infarction in past 12 months
  * Uncontrolled diabetes (HbAlc >= 7.2%) or diabetes requiring insulin injection
  * Uncontrolled hypertension (systolic >170mmHg or <90mmHg, diastolic >100mmHg or <50mmHg)
  * Immunodeficiency
  * Positive HBV, HCV, HIV, syphilis
  * pregnant or on breast feeding
  * any history of drug, alcohol abuse. mis-use
  * Any significant signs, symptoms or previous diagnosis of psychological disorder
  * Impossible to follow scheduled visits
  * Currently participating or participated in other clinical studies within past 3 months
  * Allergic to protein products (serum), antibiotics (gentamicin), DMSO (Dimethyl sulfoxide)
  * Any circumstances that is not suitable for participating or continuing clinical study or participants who clinical investigator considers not suitable for participation

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) | One month after stem cell injection
  Any TEAEs reported by patients or assessed by laboratory and image work up
Incidence of Treatment-Emergent Adverse Events | Three months after stem cell injection
  Any TEAEs reported by patients or assessed by laboratory and image work up
Incidence of Treatment-Emergent Adverse Events | Six months after stem cell injection
  Any TEAEs reported by patients or assessed by laboratory and image work up
Incidence of Treatment-Emergent Adverse Events | Nine months after stem cell injection
  Any TEAEs reported by patients or assessed by laboratory and image work up
Incidence of Treatment-Emergent Adverse Events | Twelve months after stem cell injection
  Any TEAEs reported by patients or assessed by laboratory and image work up

SECONDARY OUTCOMES:
Changes of pain after stem cell injection | Changes of Pain from baseline, 1, 3, 6, and 12 months after stem cell injection
  Assessed by VAS (Visual Analog Scale)
Changes of PUF (Pelvic Pain and Urgency/Frequency) scores after stem cell injection | Changes of PUF score from baseline, 1, 3, 6, 12 months after stem cell injection
  Assessed by PUF questionnaire
Changes of ICQ (O'Leary-Sant interstitial cystitis symptom index/problem index) scores after stem cell injection | Changes of ICQ scores from baseline, 1, 3, 6, 12 months after stem cell injection
  Assessed by ICQ questionnaire
Changes of voiding profiles after stem cell injection | Changes of voiding profiles from baseline, 1, 3, 6, 12 months after stem cell injection
  Assessed by voiding diary (frequency, nocturia, urgency, urge incontinence and mean voided volume)
Changes of Hunner lesion after stem cell injection | Changes of Hunner lesion from baseline, 1, 3, 6, 12 months after stem cell injection
  Assessed by cystoscopy (number, sized, location)

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Soo Choo, M.D, Ph.D, Principal Investigator — Professor, Asan Medical Center
Locations (1):
- Department of Urology, Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kyung YS, Hong KS, Chung HM, Hyun Shin J, Choo MS, Kim EY, Shin JM, Kang AR, Seo JW, Park J, Park SP. A single-center, phase 1/2a trial of hESC-derived mesenchymal stem cells (MR-MC-01) for safety and efficacy in interstitial cystitis patients. Stem Cells Transl Med. 2025 May 19;14(5):szaf018. doi: 10.1093/stcltm/szaf018. PMID 40387787